CLINICAL TRIAL: NCT01287728
Title: The Value of Bacterial Loads by Real Time PCR in Predicting Recurrence of Abnormal Vaginal Flora After Oral Metronidazole Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: direction de la recherche, ASSISTANCE PUBLIQUE HOPITAUX DE MARSEILLE
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-022182-10; 2010 13 (Other: AP HM)
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Abnormal Vaginal Flora

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment BY METROMIDAZOLE (Experimental)
  Interventions: Drug: Treatment BY METROMIDAZOLE

INTERVENTIONS:
Drug: Treatment BY METROMIDAZOLE — Abnormal vaginal flora (a Nugent score of 4-10 or 3 Amsel criteria) will be treated with 2g of oral metronidazole

SUMMARY:
Abnormal vaginal flora is currently diagnosed among women (20-40%). It is associated with symptoms (bad smell, vaginal discharge) and adverse out-comes in pregnant and not pregnant women. The high recurrence rate raises the long-term effectiveness of therapy. The hypothesis is the persistence of bacteria associated with vaginal flora imbalance as Atopobium vaginae and Gardnerella vaginalis. At the present time there is a lack of an accurate marker for the risk of recurrence.

DETAILED DESCRIPTION:
Women with symptomatic abnormal vaginal flora (a Nugent score of 4-10 or sup or egal 3 Amsel criteria) will be enrolled. Abnormal vaginal flora will be treated with 2g of oral metronidazole. Follow-up will be performed at 1 week,1 month and 12 months after treatment. Vaginal samples will be tested by quantitative real time PCR to determine the vaginal concentrations of A. vaginae, G. vaginalis, and Lactobacillus spp.

ELIGIBILITY:
Inclusion Criteria:

* Woman of more than 18 years, presenting vulvo-vaginal symptoms to type(chap) of smell or abnormal vaginal losses the day of the inclusion and having an imbalance of the vaginal flora objectivized by:
* The presence of at least 3 clinical criteria of Amsel ( 41 ) is a score of Nugent > 4 ( 42 )
* Woman in genital encircled period of activity (negative pregnancy test in the inclusion) and under effective contraception, including an intra-uterine device (mechanical, hormonal).
* Woman ménopausée with or without hormonal treatment (by way oral, transcutaneous, sous cutaneous, vaginal).
* Woman encircled at the time of the inclusion.
* Having Woman was treated(handled) for a vaginal infection or one imbalance of the vaginal flora more than 7 days ago.
* Woman having understood(included) the progress and the objectives of the study and having agreed to sign a lit(enlightened) consent.
* Only the profitable women of a national insurance scheme will be included

Exclusion Criteria:

* Woman presenting a sexually transmitted infection (infection with gonococcus, with Chlamydia trachomatis, with Trichomonas vaginalis) revealing on the takings realized during the consultation of inclusion but the bacteriological results(profits) of which will be known only secondarily.
* Pregnant Woman presenting to the consultation of inclusion of métrorragies either a break of the pocket of waters or an infectious complication of the pregnancy.
* Woman removing her consent during the study.
* Lost sight Woman.
* Woman deprived of freedom, judicial or administrative;
* Woman hospitalized for quite other reason that looks for her(it);
* Woman hospitalized in a sanitary establishment or social in the other purposes that the research;
* Major Woman except state to express its consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To access the value of A. vaginae and G. vaginalis loads in predicting recurrence of abnormal vaginal flora over the course of 12 months after oral metronidazole therapy. | 2 YEARS

SECONDARY OUTCOMES:
Inform the predictive and technical characteristics (sensibility and specificity) vaginal microbial concentrations | 2 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France